CLINICAL TRIAL: NCT00783341
Title: An Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of GAP-134 Administered Intravenously as 6-Day Continuous Infusions to Healthy Subjects
Brief Title: Study of the Safety, Tolerability, and Pharmacokinetics of GAP-134 Administered Intravenously
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3205K2-1001
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — 1-(2-aminoacetyl)-4-benzamidopyrrolidine-2-carboxylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GAP-134 (Experimental)
  Interventions: Drug: GAP-134
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GAP-134
  Arms: GAP-134
Drug: placebo
  Arms: placebo

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics (PK) of ascending doses of GAP 134 administered as 6-day continuous IV infusions to healthy subjects.

ELIGIBILITY:
Inclusion

1. Men or women of non childbearing potential (WONCBP) aged 18 to 50 years inclusive at screening.
2. Body mass index (BMI) in the range of 18.0 to 30.0 kg/m2 and body weight ≥50 kg.
3. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital sign measurements, and 12-lead electrocardiogram (ECG).
4. Serum creatinine level must be less than 1.30 mg/dL. (Normal range: 0.44 to 1.24 mg/dL.)
5. Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.

Exclusion

1. Presence or history of any disorder that may prevent the successful completion of the study.
2. Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
3. Any surgical or medical condition that may interfere with the distribution, metabolism, or excretion of the test article.
4. Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days before study day 1.
5. Any history of clinically important cardiac arrhythmias.
6. Familial history of long QT syndrome or unexpected cardiac death.
7. History of drug abuse within 1 year before study day 1.
8. History of alcoholism within 1 year before study day 1.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety as determined by reported adverse events, laboratory test results, and ECGs | 3 weeks

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Philadelphia, Pennsylvania, United States